CLINICAL TRIAL: NCT06984263
Title: Male Lichen Sclerosus - Risk Factors, Treatment, and Impact on Quality of Life
Status: Recruiting | Type: Observational
Sponsor: Region Västerbotten (Other Government)
Collaborators: Umeå University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-03331-01
Record Dates: First submitted 2025-05-09; First posted 2025-05-22 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Lichen Sclerosus
Keywords: lichen sclerosus
MeSH Terms: conditions — Lichen Sclerosus et Atrophicus | interventions — Circumcision, Male

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Foreskin tissue, urine, feces, and swab samples from the genital area will be collected at baseline from a subset of patients undergoing circumcision. These biospecimens will be stored for future exploratory analyses, including microbiome profiling and metabolomic analysis, with the aim of investigating potential disease mechanisms and biomarkers associated with lichen sclerosus.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- LS Urology: Male patients (≥18 years), undergoing circumcision due to phimosis at the Department of Urology. Diagnosis of lichen sclerosus (LS) confirmed by histopathological examination of the foreskin. Participants will complete questionnaires and provide biological samples (e.g., skin, urine, and fecal samples) for exploratory analyses. Follow-up will be conducted to assess long-term treatment outcomes.
  Interventions: Procedure: Circumcision
- LS dermatology: Male patients (≥18 years), diagnosed with LS in outpatient care at the Department of Dermatology. Participants will complete questionnaires and be followed over time to evaluate treatment and quality of life.
- Controls - Urology: Male patients (≥18 years), undergoing circumcision at the Department of Urology, with no histopathological evidence of LS. These participants will provide biological samples at baseline and serve as urology-based controls for comparison with LS patients.
  Interventions: Procedure: Circumcision
- Controls - General Population: Male participants (≥18 years) without any known genital symptoms or history of LS, recruited from the general population. They will complete the same questionnaire as other study groups but will not be sampled or followed longitudinally.

INTERVENTIONS:
Procedure: Circumcision — Circumcision performed as part of standard clinical care in patients with phimosis, which may be caused by lichen sclerosus. The procedure is not assigned by the study but observed as part of routine treatment
  Groups: Controls - Urology; LS Urology

SUMMARY:
This observational study aims to evaluate routine treatment outcomes in men with lichen sclerosus (LS), including a long-term follow-up to assess disease progression and histopathological changes. The study also investigates potential risk factors for LS and the disease's impact on quality of life and sexual health.

DETAILED DESCRIPTION:
Lichen sclerosus (LS) is a chronic inflammatory and scarring dermatosis with a predilection for the anogenital area. While both sexes can be affected, this study focuses on men, in whom LS can cause phimosis and may require circumcision. Topical corticosteroids are first-line treatment, but there is a lack of long-term studies evaluating the efficacy of circumcision in male LS. In addition, risk factors and the impact of LS on quality of life and sexual health are insufficiently studied.

This observational cohort study aims to follow male patients with LS over time to assess treatment outcomes, disease progression, and the potential development of epithelial atypia. Patients aged 18 years or older, Swedish-speaking, and diagnosed with LS will be recruited from both the urology and dermatology departments in Västerbotten County, Sweden. At the urology department, patients undergoing circumcision for phimosis will be included; at the dermatology department, all men diagnosed with LS will be invited to participate. All participants will provide written informed consent and will receive treatment according to standard clinical routines and national or international guidelines.

Participants will complete a standardized questionnaire regarding symptoms, quality of life, and sexual health. A control group of age-matched, Swedish-speaking men without genital symptoms will also complete the same questionnaire once but will not be followed longitudinally. For exploratory analyses, patients recruited from the urology department will also provide biological samples (e.g. foreskin, urine, feces) at baseline to facilitate future investigations of microbiome composition and metabolic profiles.

ELIGIBILITY:
Inclusion Criteria for patients with LS (LS Urology and LS dermatology):

* Biologically male
* ≥18 years old
* Referred to the dermatology department or the urology department in Västerbotten and diagnosed with LS.
* Must be able to read and write Swedish to fill in questionnaire and informed consent.

Inclusion criteria for control group "Controls - Urology":

* Biologically male
* ≥18 years old
* Phimosis without LS, treated with circumcision at the urology department in Västerbotten
* Must be able to read and write Swedish to fill in questionnaire and informed consent.

Inclusion criteria for control group "Controls - General Population":

* Biologically male with male genitalia
* ≥18 years old
* No genital symptoms
* Must be able to read and write Swedish to fill in questionnaire and informed consent.

Exclusion Criteria for all groups:

* Age under 18 years old
* Not able to read and write in Swedish.
* Unable to leave an informed consent to participate.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study includes adult men (≥18 years old), Swedish-speaking, recruited from the dermatology and urology departments in Västerbotten County, Sweden. Participants with a clinical diagnosis of lichen sclerosus (LS) will be recruited from both departments. From the urology department, additional participants undergoing circumcision for phimosis will be included; this group may include both patients with and without LS, as confirmed by histopathological examination of the foreskin. An age-matched control group of men without genital symptoms will also be included. All participants must be able to provide informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-10-06 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2038-10 (Estimated)

PRIMARY OUTCOMES:
Long-term clinical outcome of treatment for lichen sclerosus | baseline, 1 year, 3 years, 5 years, 10 years
  Assessment of symptom resolution, recurrence, and need for additional treatment over a follow-up period of up to 10 years, based on clinical assessment and patient-reported outcomes. The severity of the disease will be graded on a four point scale 0-3 (0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms, 3 = severe symptoms)

SECONDARY OUTCOMES:
Detection of epithelial atypia or dysplasia | At time of surgery and at follow-up (up to 10 years)
  Histopathological analysis of foreskin tissue obtained during circumcision to determine prevalence and incidence of epithelial atypia or dysplasia. Biopsies will be performed on clinical suspicion of cell atypia at follow-up.
Quality of life assessed by Dermatology Life Quality Index (DLQI) | Baseline, 1 year, 3 years, 5 years, 10 years. Controls assessed at baseline only
  Quality of life will be evaluated using the DLQI questionnaire. Scores range from 0 (no impact) to 30 (maximum impact).
Exploratory analysis of microbiome composition | Baseline only
  Microbiome composition will be explored using biological samples collected at baseline, including swabs from the foreskin and rectum, and urine samples. The specific sample types to be analyzed will be determined based on sample quality and feasibility. The aim is to investigate potential associations between microbial composition and LS.
Exploratory analysis of metabolomic profiles | Baseline only
  Metabolic profiles will be analyzed in selected biological samples collected at baseline (e.g., urine, foreskin tissue, and blood) from patients with LS and controls. The specific sample types to be analyzed will be determined based on sample quality and analytical feasibility. The aim is to identify metabolic signatures potentially linked to disease mechanisms.

CONTACTS AND LOCATIONS:
Locations (1):
- Umeå University Hospital, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Data on group level will be shared upon request. Sharing individual participant data must be investigated to make sure it is compliant with Swedish laws and EU regulations.